CLINICAL TRIAL: NCT04641442
Title: A Three-period Multicenter Study, With a Randomized-withdrawal, Double-blind, Placebo-controlled Design to Evaluate the Clinical Efficacy, Safety and Tolerability of MAS825 in Patients With Monogenic IL-18 Driven Autoinflammatory Diseases, Including NLRC4-GOF, XIAP Deficiency, or CDC42 Mutations
Brief Title: Study to Evaluate the Efficacy, Safety and Tolerability of MAS825 in Patients With Monogenic IL-18 Driven Autoinflammatory Diseases, Including NLRC4-GOF, XIAP Deficiency, or CDC42 Mutations
Acronym: MASter-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMAS825D12201
Record Dates: First submitted 2020-11-20; First posted 2020-11-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: NLRC4-GOF, AIFEC (Autoinflammation With Infantile Enterocolitis), XIAP Deficiency, CDC42 Mutations
Keywords: NLRC4-GOF; AIFEC; enterocolitis; autoinflammation; MAS; NLRC4 (SCAN4); XIAP deficiency; CDC42 mutations
MeSH Terms: conditions — Lymphoproliferative Syndrome, X-Linked, 2; Enterocolitis

STUDY DESIGN:
Intervention Model Description: This study includes:
  * Screening
  * Period 1: Open-Label Treatment Period to identify responders to MAS825
  * Period 2: Randomized Withdrawal Period consists of a randomized treatment withdrawal period to primarily assess the efficacy of MAS825 compared to placebo.
  * Period 3: Open-Label, Long-Term Safety follow-up
  * Period 3s: Open-Label, transition to new route of administration and safety follow-up
  * End of Study
  Patients will participate in all 3 periods of the study if they have never been treated with MAS825 before.
  Patients who are enrolled from the Managed Access program will participate in Period 3 and Period 3s only after completing screening and baseline assessments.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subject, investigator, and sponsor blinding via manual randomization during Period 2, Randomized Withdrawal Period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAS825 (Experimental): Experimental drug
  Interventions: Biological: MAS825
- Placebo (Placebo Comparator): matching placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MAS825 — Experimental drug
  Arms: MAS825
Biological: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
This study is a Phase 2 trial designed to evaluate the clinical efficacy, safety, and tolerability of MAS825 in patients with NLRC4-GOF, XIAP deficiency, or CDC42 mutations.

DETAILED DESCRIPTION:
This is a three-period study, with an open-label, single-arm active treatment in Period 1 followed by a randomized-withdrawal, double-blinded, placebo-controlled design in Period 2, and an open label, long-term safety follow-up in Period 3 and Period 3s. The total study duration is approximately 4 - 5 years.

Patients who enter Period 2 will be randomized to MAS825 or matching placebo in a 1:1 ratio.

Cohort 1 patients will complete all periods of the study, which will take approximately 5 years.

Cohort 2: Patients who are receiving MAS825 in a Novartis Managed Access Program with a diagnosis of NLRC4-GOF, XIAP deficiency, or CDC42 mutation who meet criteria will be eligible to directly enter into Period 3 and Period 3s for open-label long-term safety follow-up. Cohort 2 patients will be in the study for approximately 4 years.

ELIGIBILITY:
Inclusion Criteria:

For all Patients:

1. Male and female patients weighing at least 3 kg
2. Written informed consent by parent(s)/legal guardian(s) for the pediatric patients and assent by the pediatric patient (depending on local requirements) must be obtained before any study-specific assessment is performed. For adult patients, written informed consent by patients capable of giving consent, or when the patient is not capable of giving consent, by his/her legal/authorized representative (if allowed according to local requirements).

   Cohort 1 specific inclusion criteria:
3. Patients with a genetic diagnosis of either NLRC4-GOF, XIAP deficiency, or CDC42 mutation
4. Clinical history and investigations consistent with autoinflammation and infantile enterocolitis (AIFEC/NLRC4-GOF), XIAP or CDC42. XIAP patients must have persistent disease or be resistant to escalating therapy.
5. At first treatment, evidence of active disease as assessed by inflammatory markers and PGA

   Cohort 2 specific inclusion criteria:
6. Patients with a genetic diagnosis of NLRC4-GOF, XIAP deficiency, or CDC42 mutations who are being treated with MAS825 in a Novartis Managed Access Program (MAP).

Exclusion Criteria:

1. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes or to any of the excipients.
2. Signs and symptoms, in the judgment of the investigator, of clinically significant active bacterial, fungal, parasitic or viral infections, excluding chronic Epstein-Barr Virus (EBV).

   - COVID-19 specific: If in line with health and governmental authority guidance, it is highly recommended that testing to exclude COVID-19 using PCR or comparable approved methodology be completed within 1 week prior to first dosing.
3. Any conditions or significant medical problems, which in the opinion of the investigator places the patient at unacceptable risk for MAS825 therapy
4. Previous treatment with anti-rejection and/or immunomodulatory drugs within the past 28 days or 5 half-lives (whichever is the longer) for immunomodulatory therapeutic antibodies (or as listed in the prohibited medications section) prior to MAS825 treatment with the exceptions of glucocorticoids, cyclosporin and targeted binding or blocking therapies.
5. A positive HIV test result at Screening. Evidence of prior testing within 3 months is sufficient.
6. A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result at Screening. Evidence of prior testing within 3 months is sufficient.
7. Presence of tuberculosis infection as defined by a positive TB test at Screening. Evidence of prior testing within 3 months is sufficient.
8. Live vaccinations within 1 month prior to MAS825 treatment, during the trial, and up to 3 months following the last dose.
9. Pregnant or nursing (lactating) females.
10. Female patients of child-bearing potential (or Tanner stage 2 or above) who are or might become sexually active, agree to use highly effective contraceptive methods to prevent pregnancy while on MAS825 therapy
11. Patients weighing >160 kg at Screening.
12. For CDC42 mutation patients: Takenouchi-Kosaki syndrome - CDC42 mutations associated with a diverse syndrome characterized by variable development delays, cardiac, brain and hematological abnormalities.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Occurrence of disease flare in patients with MAS825 treated patients compared with placebo during Period 2 assessed by Physician's Global Assessment and inflammatory markers | Period 2
  To determine the efficacy of MAS825 in prevention of flares in patients with monogenic IL-18 driven autoinflammatory diseases, including NLRC4-GOF, XIAP deficiency or CDC42 mutations

SECONDARY OUTCOMES:
All cohorts: Number and severity of safety assessments and adverse events | Screening through EOS (End of Study)
  To evaluate the safety and tolerability of MAS825
All cohorts: Confirmation of serological markers of MAS825 | Day 1 through EOS
  Evaluate the serological markers of MAS825
Cohort 1: PGA and inflammatory markers | Day 29, end of Period 1, end of Period 2
  Evaluate the efficacy of MAS825 to improve the clinical status of patients with NLRC4-GOF, XIAP deficiency or CDC42 mutations
Cohort 1: Serological remission via inflammatory markers | Day 29, end of Period 1, and end of Period 2
  Evaluate efficacy of MAS825 to achieve serological remission
Cohort 1: Glucocorticoid therapy <0.2mg/kg by end of period 1 | End of Period 1
  Evaluate the effect of MAS825 on concomitant glucocorticoid administration
Cohort 1: Time to first flare | Period 2
  Evaluate effect of MAS825 on the time to first flare
All cohorts: Physician Severity Assessment of Disease Signs and Symptoms scale | Screening through EOS
  Evaluate the efficacy of MAS825 to improve signs and symptoms of the disease
All cohorts: Patient / Parent global assessment of disease activity (PPGA) scale | Screening through EOS
  Evaluate effect of MAS825 on patient reported outcomes over time

CONTACTS AND LOCATIONS:
Locations (19):
- United States (8):
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children´s Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Childrens Hospital, Houston, Texas
  - Texas Children´s Hospital, Houston, Texas
  - Seattle Childrens Hospital, Seattle, Washington
  - Seattle Children´s Hospital, Seattle, Washington
- Czechia (3):
  - Centrum detske revmatologie a autoinflamatornich onemocneni, Prague, CZ
  - Novartis Investigative Site, Prague
  - Ustav Imunologie 2 LF UK a FN Motol, Prague
- Novartis Investigative Site, Paris, France
- Italy (2):
  - Bambino Gesu Hospital, Roma, RM
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Chiba, Japan
- Spain (2):
  - Hospital Clinic Barcelona, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com